CLINICAL TRIAL: NCT03300323
Title: The Impact of Different Rates of Administration of a Fluid Challenge on the Proportion of Responders and Non-responders in the Post-operative Patient
Brief Title: Response to Varying the Rate of Administration of a Fluid Challenge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St George's Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 17.0092
Record Dates: First submitted 2017-09-14; First posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Peri-operative Fluid Management
Keywords: peri-operative; fluid; microcirculation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV Fluid challenge administration _5 (Active Comparator): 4ml/kg intravenous fluid challenge administered over 5 minutes
  Interventions: Diagnostic Test: IV fluid challenge administration
- IV Fluid challenge administration 20 (Active Comparator): 4ml/kg intravenous fluid challenge administered over 20 minutes
  Interventions: Diagnostic Test: IV fluid challenge administration

INTERVENTIONS:
Diagnostic Test: IV fluid challenge administration — Administration of an intravenous fluid challenge to assess for fluid responsiveness

SUMMARY:
Administration of intravenous fluids is a key step in the management of the post-operative patient. Fluid management has been identified as one area that can affect rates of post-operative complications and outcomes. It is important to give the right amount of fluid, enough to optimise cardiovascular function, but not so much that we flood the cells. To guide this, we use a fluid challenge, administration of a small amount of fluid to test the cardiovascular response. At present there is significant inter-user variability in the method of administration of a fluid challenge. To ensure accuracy and reliability in assessing the response to a fluid challenge, the optimal method of administration needs to be determined.

The aim of this study is to investigate the optimal rate to give a fluid challenge over. Patients will be randomised to receive a fluid challenge over either 5 or 20 minutes. Both of these rates are within the currently accepted range. All patients will receive a dose of 4ml/kg of intravenous fluid. Previous work has shown this to be the optimal dose to reliably stress the system.

Measurement of the mean pressure in the cardiovascular system (mean systemic filling pressure or Pmsf) during the administration of a fluid challenge will be used to assess which rate of administration effectively challenges the cardiovascular system. Pmsf is measured using a pneumatic tourniquet inflated for sixty seconds, above an arterial line. The invasive arterial pressure is observed to then determine Pmsf. Cardiac output will also be monitored during and after administration of the fluid challenge. Since the microcirculation may remain impaired despite stabilisation of the macrocirculation, we will also observe this at baseline, on completion of the fluid challenge, and at 5 minute intervals for 15 minutes. This is observed using a handheld camera placed under the tongue.

The hypothesis is that administration of a fluid challenge at a faster rate, over 5 minutes as opposed to 20 minutes, will be a more effective test of the cardiovascular response. An effective fluid challenge is defined as one that causes a significant rise in mean systemic filling pressure. As such, a higher proportion of responders will be seen in response to the faster rate of fluid challenge. A responder is defined by an increase in cardiac output or stroke volume of more than 10% from baseline in response to a fluid challenge.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgical patients admitted post-operatively to the General and Cardiothoracic Intensive Care Unit, requiring optimization with fluid therapy, as per the current clinical indications.
* Adult patients, aged >18 years, who have given informed consent to participate in the study.

Exclusion Criteria:

* Patients without capacity to consent for themselves
* Patients requiring aggressive fluid resuscitation due to life-threatening cardiovascular instability, such would not allow for period of observation for stability as defined in protocol.
* Pregnancy
* Possible contraindications to the use of the cardiac output monitoring device, or pathology known to affect accuracy of readings, including

  * Extensive peripheral arterial occlusive disease in upper limbs
  * Postoperative valvular insufficiency
  * New onset arrhythmia
  * Cardiac assist device
  * Right ventricular failure, (formal pre-operative diagnosis)
  * Severe left ventricular failure or diastolic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Clinical response to fluid administration - SV and/or CO response | 35 minutes
  A response is defined by an increase in SV and/or CO by more than 10% from the starting point of fluid administration Patients are randomised to two groups and administrated fluid at two different rates. The proportions of responders in the two groups are compared.

SECONDARY OUTCOMES:
Pharmacodynamic response to fluid administration - mean systemic filling pressure (Pmsf) | 35 minutes
  The pharmacodynamic response to fluids, in terms of maximum change and duration of change in Pmsf with different rates of fluid administration.
Pharmacodynamic response to fluid administration - cardiac output | 35 minutes
  The pharmacodynamic response to fluids, in terms of maximum change and duration of change in CO with different rates of fluid administration.
Pharmacodynamic response to fluid administration - blood pressure | 35 minutes
  The pharmacodynamic response to fluids, in terms of maximum change and duration of change in arterial blood pressure with different rates of fluid administration.
Microcirculation | 35 minutes
  The response seen within the microcirculation with varying the rate of administration of the fluid challenge.

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Cecconi, Study Chair — St George's University Hospital

IPD SHARING:
Plan to Share IPD: No